CLINICAL TRIAL: NCT03772015
Title: The Change in Vaginal Axis on MRI After Uterus Preserving Laparoscopic Lateral Mesh Suspension
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Collaborators: Bartin State Hospital (Other Government)
Responsible Party: Principal Investigator, OZAN DOGAN, Principal Investigator, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 240918
Record Dates: First submitted 2018-12-09; First posted 2018-12-11 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Prolapse Genital; Anatomical Pathological Condition
Keywords: laparoscopic lateral mesh suspension; lateral abdominocervicopexy; apical prolapse; anterior prolapse; vaginal axis; magnetic resonance imaging
MeSH Terms: conditions — Pathological Conditions, Anatomical | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study: Patients who had the operation of "laparoscopic lateral mesh suspension" for apical prolapse will have magnetic resonance imaging preoperatively and at postoperative 6th month
  Interventions: Diagnostic Test: Magnetic resonance imaging
- Control: Multiparous, sexually active participants who have grade 0 or 1 (asymptomatic if exists) prolapse will have magnetic resonance imaging as a control group
  Interventions: Diagnostic Test: Magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: Magnetic resonance imaging — MRI will be performed using a standard body spiral in the supine position with 5 mm section thickness, on the axial, coronal and sagittal planes and the diffusion weighted images acquired will be evaluated by a specialised radiologist who will be blind to the participants.

SUMMARY:
Laparoscopic lateral mesh suspension is emerged as a practical, safe and feasible alternative to sacropexy to treat female genital apical prolapse. Investigators hypothesized that uterus-preserving lateral suspension provides a better anatomical positioning.

DETAILED DESCRIPTION:
Suspending the cervix to the bilateral abdominal wall through subperitoneal tunnels may properly mimic cardinal ligament and restore the normal vaginal axis. To prove the null hypothesis, it is planned to compare the vaginal axis on Magnetic Resonans Imaging taken preoperatively and postoperatively in patients who are scheduled for lateral mesh suspension for apical prolapse.

ELIGIBILITY:
Inclusion Criteria:

* Female genital prolapse

Exclusion Criteria:

* Patients who had pouch of Douglas obliteration
* Patients with enterocele
* Patients who have any congenital or acquired anatomic and reproductive anomaly

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled for lateral mesh suspension operation to treat apical prolapse.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2018-12-09 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Vaginal axis | at 6th months after the operation
  From the images obtained in the sagittal plane, the vagina, which will be observed as a high signal intensity linear structure in T2A images, and the levator plate extending as a flow-signal intensity flat structure in T1A images, will be evaluated.
  The angles between the pubococcygeal line and lower vaginal segment (angle A), between the levator plate and the pubococcygeal (angle B) and between lower and upper vaginal segments (angle C) will be measured.
Vaginal distances | at 6th months after the operation
  The distance between the posterior vaginal fornix and the midpoint of the anterior side of the 2nd vertebra will be measured in the mid-sagittal plane (PF-S2). The distance between the right spina ischiadica and right vaginal fornix (RSI-RF), and, the distance between the left spina ischiadica and left vaginal fornix (LSI-LF) will be measured on T2A images acquired in the axial plane.

SECONDARY OUTCOMES:
Urge Symptoms | Evaluation at postoperative 6th month
  Michigan Incontinence Severity Index (M-ISI) scale will be used to assess subjective outcome including urge symptoms. This scale has ten items, consisting of a total M-ISI domain (the sum of items 1-8) and a distinct Bother domain (the sum of items 9 and 10). The total M-ISI score consists of three subdomains (items 1-3 for stress urinary incontinence [SUI], items 4-6 for urge urinary incontinence [UUI], and items 7 and 8 for Pad usage [PU]. The responses for each item range from 0 to 4 on a Likert-type scale, with higher values representing greater symptoms and greater bother. Total domain and subdomain scores are obtained by simply adding the respective answers. The minimally important difference has been determined for the following domains/subdomains: total M-ISI (4 points), SUI (2 points), UUI (2 points), and PU (1 point).
Prolapse symptoms | Evaluation at postoperative 6th month
  The POP-SS consists of seven items, each with a 5-point Likert response set (0 = never, 1 = occasionally, 2 = sometimes, 3 = most of the time and 4 = all of the time). A total score (range 0-28) is calculated by summing the seven individual symptom responses to derive the POP-SS score. In addition, women indicate which one of the seven symptoms causes them most bother.
Sexual functions | Evaluation at postoperative 6th month
  The FSFI evaluates sexual functioning in women and comprises of 19 questions with different answer choice scales referring the sexual life in the previous 4 weeks. The answer choices in the FSFI carry a number of points and are summed to obtain six domain scores and an overall score. For the latter, there is a threshold at 26.55 which means tFhat all values below are classed as indicating female sexual dysfunction (FSD). The domain scores are obtained as the sum of points attributed to questions in that domain multiplied by the domain factor.

CONTACTS AND LOCATIONS:
Overall Officials: Ozan Dogan, MD, Principal Investigator — Hamidiye Sisli Etfal Training and Research Hospital; Murat Yassa, MD, Principal Investigator — Bartin State Hospital
Locations (1):
- Hamidiye Sisli Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Senturk MB, Kilicci C, Aydin S, Polat M, Abide Yayla C, Karateke A. Vaginal axis on MRI after unilateral and bilateral sacral hysteropexy: a controlled study. J Obstet Gynaecol. 2018 Jan;38(1):115-120. doi: 10.1080/01443615.2017.1336754. Epub 2017 Aug 17. PMID 28816554